CLINICAL TRIAL: NCT02278224
Title: Rumination Focused Cognitive Behavioral Therapy for Major Depression and Recurrent Depression and Relapse Prevention -a Pragmatic RCT Study in a Danish Psychiatric Outpatient Service
Brief Title: Rumination Focused Cognitive Behavioral Therapy for Major Depression and Recurrent Depression
Acronym: RuCoD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Exeter (Other); The University of Western Australia (Other)
Responsible Party: Principal Investigator, Morten Hvenegaard, Cand.psych. Ph.d. student, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RuCoD-CPH; RuCoD-UoC (Other: University of Copenhagen)
Record Dates: First submitted 2014-08-31; First posted 2014-10-29 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Depression; Recurrent Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rumination Focused CBT (Experimental): 11 sessions of manualised group based Rumination Focused CBT for depression. 3 hours sessions are administered once during 11 weeks in groups of approximately 8 patients and two therapist.
  Interventions: Behavioral: Group based rumination focused CBT
- Cognitive Behavioral Therapy (Active Comparator): 11 sessions of manualised group based CBT for depression. 3 hours sessions are administered once during 11 weeks in groups of approximately 8 patients and two therapist.
  Interventions: Behavioral: Group based CBT

INTERVENTIONS:
Behavioral: Group based rumination focused CBT — The RFCBT is a group trans-diagnostic manual based psychotherapy for depression and anxiety. RFCBT focuses on increasing effective behaviour - i.e., not stopping rumination but making it functional. It's grounded within the core principles and techniques of CBT for depression with two adaptations: (1) a functional-analytical perspective using Behavioural Activation (BA) approaches, (2) an explicit focus on shifting processing style via imagery and experiential approaches.
  Arms: Rumination Focused CBT
Behavioral: Group based CBT — The control group is gold standard group based CBT based on Becks manual for CBT for depression.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
Group based cognitive behavioural therapy (CBT) is an effective treatment of depression, however, one third of patients do not respond satisfactorily (McDermut, Miller, & Brown, 2001), and relapse rates around 30% have been reported from several studies (Butler, Chapman, Forman, & Beck, 2006).

The present study compares group based CBT with rumination focused CBT for depression with respect to outcome and relapse.

Rumination has been evidenced as a crucial vulnerability to depression (Smith & Alloy, 2009), predicting the onset, severity and duration of future depression (Nolen-Hoeksema, 2000). Depressed individuals show a negative bias in the perception of facial emotion, in the acute phase as well as in remission (Bouhuys, Geerts, & Gordijn, 1999), and display difficulties in disengaging from negative stimuli (Koster, De Raedt, Goeleven, Franck, & Crombez, 2005). In addition the present study investigate rumination and perceptual attention bias as potential key mechanisms underlying depression.

128 depressed patients will be recruited and randomised for group based CBT or group based rumination focused CBT. Patients are assessed subsequently during treatment and at 6 month follow-up regarding depression, rumination, worry, negative perceptual bias, attention control. Results are expected at spring 2016.

DETAILED DESCRIPTION:
Background and rationale

The aim of the present study is to compare the effectiveness of rumination-focused cognitive behavior therapy vs. cognitive behavior therapy for treatment of depression.

Understanding the mechanisms involved in effective cognitive behavioural therapy is a key focus of clinical research (Watkins, 2009). The study will investigate possible underlying mechanisms of rumination and thereby provide insights about the information processing and symptoms of depression.

Rumination, a process of recurrent negative thinking and dwelling on negative affect, is a common residual symptom (Kim, Yu, Lee, & Kim, 2012; Riso et al., 2003). Rumination has been evidenced as a crucial vulnerability to depression (Smith & Alloy, 2009), predicting the onset, severity and duration of future depression (Nolen-Hoeksema, 2000).

Such knowledge indicates that rumination is a key factor involved in the initiation and maintenance of depressive symptoms. Individuals that display high levels of rumination even if not currently presenting depressive symptoms may therefore have an increased risk for developing future depression. Consequently, if involved in the pathogenesis of depression, rumination may constitute an active ingredient of psychological intervention. Hence, interventions explicitly targeting rumination may improve the efficiency of CBT for recurrent and chronic depression (Watkins, 2009). However, few studies have tested interventions targeting rumination, with the exception of Watkins (2007; 2011).

Cognitive theories argue that information processing bias influences the aetiology and maintenance of depression. On tests of cognitive performance, particularly attention and memory has been repeatedly reported affected in depression (Goeleven, De Raedt, Baert, & Koster, 2006). Depressed individuals show a negative bias in the perception of facial emotion, in the acute phase as well as in remission (Bouhuys, Geerts, & Gordijn, 1999), and display difficulties in disengaging from negative stimuli (Koster, De Raedt, Goeleven, Franck, & Crombez, 2005).

It is suggested in the literature that depressed people are not able to gain control over the emotional influence of negative stimuli due to dysfunctional inhibition of negative stimuli (Donaldson, Lam, & Mathews, 2007). This idea is substantiated by the strong relationship between rumination and depression suggesting that impaired inhibitory function may be an underlying mechanism of rumination.

However, experimental paradigms used to study attention has, apart from Donaldson and colleagues (2007), not been applied to rumination or other self-report measures assessing attention and attentional control in clinical samples. The present study investigates the relationship between clinical features of depression such as the self-reported tendency to ruminate in response to negative affect, as well as the experience of attentional control and actual performance on cognitive tests assessing attentional control. Furthermore by combining clinical self-report with test performance, the study addresses potentially underlying mechanisms of rumination. Understanding the mechanisms involved in effective cognitive behavioural therapy is thus a key focus of clinical research (Watkins, 2009).

RFCBT will be compared to CBT for depression. Cognitive Behavioural Therapy (CBT) is recommended for the treatment of depression by the National Institute for Health and Clinical Excellence (NICE) in UK. Group CBT is an effective treatment of depression, however, one third of patients do not respond satisfactorily (McDermut, Miller, & Brown, 2001), and relapse rates around 30% have been reported from several studies (Butler, Chapman, Forman, & Beck, 2006). Residual symptoms following treatment is a common problem, as 30-50% of remitted patients present residual symptoms by the end of treatment (Kennedy & Paykel, 2004). These patients display more depressive symptoms, have a lower level of social functioning and utilize more health care services (Cornwall & Scott, 1997) compared to fully remitted patients.

Objectives:

The aim of the present study to compare the effectiveness of rumination-focused CBT vs. CBT for treatment of depression.

Trial design:

The design is a pragmatic block randomized controlled blinded trial comparing two types of group based cognitive behavioural therapy for depression.

Study design:

The study takes place in a community psychiatric outpatient service in Hillerød, Denmark, which receives 200-250 patients with depression per year. Patients that are referred for treatment at the Psychiatric Outpatient Centre in Hillerød with a primary diagnosis of depression, recurrent or chronic, are recruited to the study. We plan to recruit a total of 128 patients, 64 in each treatment type. Intake will take place from July 2013 until Marts 2015.

Therapists conducting the group therapies are trained and experienced cognitive behavioural therapist with at least 4 years of experience with CBT. The therapist conduction the groups with RFCBT are trained and supervised by professor Ed Watkins (affiliation).

Both interventions runs for 11 week with a 3 hours session once a week and will be delivered by trained clinicians with at least two years of experience in CBT. Preceding the first group session the participants will be given an individual session with a group therapist to prepare for the groupbased treatment.

The psychiatrist conducting the initial evaluation of the patients invites the patients to participate if the inclusion criteria are met. The patients will receive verbal and written information about the project from the psychiatrist. If interested in participation the patients will be contacted by the Ph.D. student to sign the informed consent and invited to first assessment. After the assessment the patients are finally randomised by computer method to receive one of the two treatment types.

Primary outcome:

Primary outcome is the post-treatment assessment of the Hamilton Rating Scale for Depression (HRSD) Bech P, Kastrup M, Rafaelsen OJ. (1986).

Secondary outcomes:

Post-treatment measures of HAM-D-6 (Bech et al., 1975), Penn State Worry Questionnaire (PSWQ; Meyer, Miller, Metzger, & Borkovec, 1990), Ruminative Response Scale of the Response Style Questionnaire (RRS;(Nolen-Hoeksema & Morrow, 1991), Generalized Anxiety Disorder 7 (GAD-7; Spitzer, et al. 2006). Trail-making A and B (Strauss et al. 2006), Dot-probe task -computerized test of cognitive control and emotional processing (Donaldson et al., 2007).

Sample size estimation:

Assuming similar mean changes in HRSD scores from pre-to-post intervention as found by Watkins and colleagues [18] for RFCBT (M = 7.81) and by Paykel and colleagues [11] for CBT (M = 3.52), and a conservative estimate of pooled standard deviation for change in HRSD of 6 (when SD= 3.60 for change in HRSD in RFCBT), we estimate a between-treatment effect size of Cohen's d = 0.7. To detect a difference in effect size of 0.7 between RFCBT and CBT at a two-tailed significance level of 5%, each treatment arm requires 44 patients each to obtain 90% statistical power [40]. Assuming a dropout rate of 20%, we will recruit 55 patients into each treatment arm. With an average size of the therapy group of m = 8 in both treatment arms, and an intraclass correlation of about ρ = 0.05, a design effect of 1 + (m - 1)ρ = 1.35 follows, so that we plan to recruit 8 groups in each treatment arm (128 patients in total).

Statistical analysis:

The primary outcome is the post-treatment score on the HRSD, which is treated as a continuous, normally distributed variable. The primary efficacy hypothesis will be tested using a multilevel two-group comparison (RFCBT vs. CBT), with Group as a main effect, Therapy Group as a random intercept, and the HRSD baseline score as a continuous covariate. The test will be performed at the 5% two-tailed significance level.

The primary test for efficacy will be based on the intention-to-treat population, with all randomized patients entering the analysis set, and multiple imputation of missing values in the primary endpoint [42]. For the secondary outcomes, similar analyses will be used, taking into consideration the scale of the variable (e.g., logistic regression for binary outcomes).

Ethical considerations:

The patients will be informed about the research project and purpose of the project prior to participation and asked for informed consent. There are no side effect due to the rumination focused cognitive behavioral therapy. It is not possible to pay the patients for the participating in the research project.

Participant can leave the treatment on request. If anyone involved in the trial get knowledge of increased risk of suicide among participants relevant prevention will be initiated.

The participant will be given treatment as usual, clinical management and medical treatment if needed assessed by highly trained psychiatrist at PCN.

The project is approved by the Danish national ethical scientific committee and is registered at The Danish Data Protection Agency by Region Hovedstaden Psychiatry (casenumber H-1-2013-049).

ELIGIBILITY:
Inclusion Criteria:

* Depression or recurrent depression with Hamilton score of 13 or above.

Exclusion Criteria:

* Bipolar disorder
* Psychotic disorder
* Substance abuse
* Eating disorder
* Functional illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2013-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale 17 | up to 6 months follow up
  The Hamilton Rating Scale for Depression (HRSD), also called the Hamilton Depression Rating Scale (HDRS), abbreviated HAM-D, is a multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery

CONTACTS AND LOCATIONS:
Overall Officials: Stig B Poulsen, Ph.d., Study Chair — University of Copenhagen
Locations (1):
- Psychiatric Outpatient Service, Hilleroed, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Cuijpers P, Karyotaki E, Weitz E, Andersson G, Hollon SD, van Straten A. The effects of psychotherapies for major depression in adults on remission, recovery and improvement: a meta-analysis. J Affect Disord. 2014 Apr;159:118-26. doi: 10.1016/j.jad.2014.02.026. Epub 2014 Feb 24. PMID 24679399
- [Background] McDermut W, Miller IW, Brown RA: The Efficacy of Group Psychotherapy for Depression: A Meta-analysis and Review of the Empirical Research. Clinical Psychology: Science and Practice 2006, 8:98-116.
- [Background] Butler AC, Chapman JE, Forman EM, Beck AT. The empirical status of cognitive-behavioral therapy: a review of meta-analyses. Clin Psychol Rev. 2006 Jan;26(1):17-31. doi: 10.1016/j.cpr.2005.07.003. Epub 2005 Sep 30. PMID 16199119
- [Background] Dimidjian S, Hollon SD, Dobson KS, Schmaling KB, Kohlenberg RJ, Addis ME, Gallop R, McGlinchey JB, Markley DK, Gollan JK, Atkins DC, Dunner DL, Jacobson NS. Randomized trial of behavioral activation, cognitive therapy, and antidepressant medication in the acute treatment of adults with major depression. J Consult Clin Psychol. 2006 Aug;74(4):658-70. doi: 10.1037/0022-006X.74.4.658. PMID 16881773
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] Kennedy N, Paykel ES. Residual symptoms at remission from depression: impact on long-term outcome. J Affect Disord. 2004 Jun;80(2-3):135-44. doi: 10.1016/S0165-0327(03)00054-5. PMID 15207926
- [Background] Riso LP, du Toit PL, Blandino JA, Penna S, Dacey S, Duin JS, Pacoe EM, Grant MM, Ulmer CS. Cognitive aspects of chronic depression. J Abnorm Psychol. 2003 Feb;112(1):72-80. PMID 12653415
- [Background] van Rijsbergen GD, Kok GD, Elgersma HJ, Hollon SD, Bockting CL. Personality and cognitive vulnerability in remitted recurrently depressed patients. J Affect Disord. 2015 Mar 1;173:97-104. doi: 10.1016/j.jad.2014.10.042. Epub 2014 Nov 4. PMID 25462402
- [Background] Vittengl JR, Clark LA, Dunn TW, Jarrett RB. Reducing relapse and recurrence in unipolar depression: a comparative meta-analysis of cognitive-behavioral therapy's effects. J Consult Clin Psychol. 2007 Jun;75(3):475-88. doi: 10.1037/0022-006X.75.3.475. PMID 17563164
- [Background] Paykel ES, Scott J, Teasdale JD, Johnson AL, Garland A, Moore R, Jenaway A, Cornwall PL, Hayhurst H, Abbott R, Pope M. Prevention of relapse in residual depression by cognitive therapy: a controlled trial. Arch Gen Psychiatry. 1999 Sep;56(9):829-35. doi: 10.1001/archpsyc.56.9.829. PMID 12884889
- [Background] Jarrett RB, Vittengl JR, Clark LA. How much cognitive therapy, for which patients, will prevent depressive relapse? J Affect Disord. 2008 Dec;111(2-3):185-92. doi: 10.1016/j.jad.2008.02.011. Epub 2008 Mar 21. PMID 18358541
- [Background] Watkins ER. Depressive rumination: investigating mechanisms to improve cognitive behavioural treatments. Cogn Behav Ther. 2009;38 Suppl 1(S1):8-14. doi: 10.1080/16506070902980695. PMID 19697180
- [Background] Watkins E, Scott J, Wingrove J, Rimes K, Bathurst N, Steiner H, Kennell-Webb S, Moulds M, Malliaris Y. Rumination-focused cognitive behaviour therapy for residual depression: a case series. Behav Res Ther. 2007 Sep;45(9):2144-54. doi: 10.1016/j.brat.2006.09.018. Epub 2007 Mar 26. PMID 17367751
- [Background] Smith JM, Alloy LB. A roadmap to rumination: a review of the definition, assessment, and conceptualization of this multifaceted construct. Clin Psychol Rev. 2009 Mar;29(2):116-28. doi: 10.1016/j.cpr.2008.10.003. Epub 2008 Nov 5. PMID 19128864
- [Background] Nolen-Hoeksema S, Wisco BE, Lyubomirsky S. Rethinking Rumination. Perspect Psychol Sci. 2008 Sep;3(5):400-24. doi: 10.1111/j.1745-6924.2008.00088.x. PMID 26158958
- [Background] Nolen-Hoeksema S. The role of rumination in depressive disorders and mixed anxiety/depressive symptoms. J Abnorm Psychol. 2000 Aug;109(3):504-11. PMID 11016119
- [Background] Watkins ER, Mullan E, Wingrove J, Rimes K, Steiner H, Bathurst N, Eastman R, Scott J. Rumination-focused cognitive-behavioural therapy for residual depression: phase II randomised controlled trial. Br J Psychiatry. 2011 Oct;199(4):317-22. doi: 10.1192/bjp.bp.110.090282. Epub 2011 Jul 21. PMID 21778171
- [Background] Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96. doi: 10.1111/j.2044-8260.1967.tb00530.x. No abstract available. PMID 6080235
- [Derived] Hvenegaard M, Moeller SB, Poulsen S, Gondan M, Grafton B, Austin SF, Kistrup M, Rosenberg NGK, Howard H, Watkins ER. Group rumination-focused cognitive-behavioural therapy (CBT) v. group CBT for depression: phase II trial. Psychol Med. 2020 Jan;50(1):11-19. doi: 10.1017/S0033291718003835. Epub 2019 Jan 11. PMID 30630555
- [Derived] Hvenegaard M, Watkins ER, Poulsen S, Rosenberg NK, Gondan M, Grafton B, Austin SF, Howard H, Moeller SB. Rumination-focused cognitive behaviour therapy vs. cognitive behaviour therapy for depression: study protocol for a randomised controlled superiority trial. Trials. 2015 Aug 11;16:344. doi: 10.1186/s13063-015-0875-y. PMID 26260780